CLINICAL TRIAL: NCT06936332
Title: A 7-week, Open Label, Single Arm Study Evaluating the Efficacy and Safety of Omnilux Clear® on Mitigating Mild to Moderate Acne in Healthy Male and Female Teenagers and Adults
Brief Title: Study Evaluating the Efficacy and Safety of Omnilux Clear on Mitigating Mild to Moderate Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablon Skin Institute Research Center (Other)
Collaborators: GlobalMed Technologies Co. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMT-OCL-01
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Acne
Keywords: acne; Light Emitting Diode Device
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Open label study evaluating the efficacy and safety
Masking Description: Open label study evaluating the efficacy and safety
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Omnilux Clear Treatment (Other): Omnilux Clear treatment of the facial area 4 times per week for 6 weeks. Total of 24 treatments.
  Interventions: Device: Omnilux Clear Light Emitting Diode Treatment

INTERVENTIONS:
Device: Omnilux Clear Light Emitting Diode Treatment — Omnilux Clear is a medical-grade, home light emitting diode (LED) treatment for acne-prone skin, using the most clinically effective LED's available, optimized for superior results. The blue light (415nm) targets and kills P. acnes bacteria living on the skin's surface. Red light (633nm) penetrates the dermis, triggering the body's own natural healing response, including the production of new collagen, the downregulation of excess oils, and the reduction of inflammation and redness.

SUMMARY:
The goal of this clinical trial is to further substantiate the effectiveness and safety of Omnilux Clear as a stand-alone treatment of mild to moderate acne in healthy teenagers and adults 14 years of age or older over the course of 7 weeks. Participants will be screened to determine eligibility, assessed, instructed on how to use the Omnilux Clear and then treated with Omnilux Clear under the direction of the study staff during the first office visit. The first treatment will also act as a photosensitivity "patch" test to evaluate the participant for any unknown hereditary photosensitivity conditions or allergies to surface contacting materials. The particpants will then treat their face with the Omnilux Clear device at home 4 times per week for the first 6 weeks of the trial. The treatments are 10 minutes in duration. Participants will return to the study site at week 3 and week 7 for assessments, photographs and questionnaires.

DETAILED DESCRIPTION:
Acne is the top skin concern for individuals in the United States. It affects subjects both physically and psychologically. While the etiology of acne is multifactorial, it does develop when the sebaceous glands in a person's skin produce excess oil. This oil combines with cells that line the gland walls and clogs the skin's pores. Normal skin bacteria (Cutibacterium acnes) colonize these pores leading to the inflammation or reddening of the skin that we associate with acne.

Increasing numbers of individuals are seeking non-invasive procedures for improving medical and aesthetic dermatologic conditions. Phototherapy refers to the use of nonthermal, noninvasive light to achieve a therapeutic outcome and can apply to a variety of light-emitting devices. Interest in recent advances in the use of light emitting diodes (LED's) have led to their clinical application for a variety of medical and cosmetic uses. Depending on the target chromophore, different wavelengths of light are used. Two wavelengths of light that have demonstrated therapeutic benefit for the treatment of acne are blue (415 nm), red (633 nm) Recent publications have reignited an interest in the numerous studies performed or sponsored by a leader in the field of LED phototherapy (Omnilux™; GlobalMed Technologies, Napa, CA) which clearly demonstrate the significant value of phototherapy for a range of clinical applications.

The option to offer non-invasive devices to all age individuals for the improvement of acne, is desirable. As oral medications have become less popular, home units that actually improve acne, with no pain and no downtime are indispensible. The benefits of light emitting diode (LED) therapy has become widely recognized in modern medicine. Benefits come from the specific wavelengths to target inflammation, bacteria, and healing tissue. Omnilux Clear® is a medical-grade, home LED treatment for acne-prone skin, using the most clinically effective LED's available, optimized for superior results. The blue light (415nm) targets and kills P. acnes bacteria living on the skin's surface. Red light (633nm) penetrates the dermis, triggering the body's own natural healing response, including the production of new collagen, the downregulation of excess oils, and the reduction of inflammation and redness. This FDA approved device not only reduces active acne and blemishes, redness and inflammation, but can help clear breakouts faster, reduce and soften the appearance of acne scarring all in a natural, painless way with no downtime.

The purpose of this open label, single-arm clinical research study is to further substantiate the efficacy and safety of Omnilux Clear® medical grade, home LED face mask treatment as a stand-alone treatment in the mitigation of mild to moderate acne in thirty (30) healthy male and female subjects, 14 years of age or older over the course of seven (7) weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or females of all Fitzpatrick Skin Types who are 14 years of age or older.
2. Subjects must be willing to provide verbal understanding and sign an Informed Consent Form, HIPAA Form and Photography Release Form approved by the Institutional Review Board. Subjects less than age of consent must sign an assent for the study and a parent must sign the informed consent (if subject reaches the age of consent during the study they should be re-consented at the next study visit).
3. Subjects must be in general good health, as determined by the Investigator.
4. Subjects willing to undergo a brief physical exam to include height, weight, blood pressure, pulse, and basic systems evaluation (Skin, Respiratory, Cardiovascular, Gastrointestinal, Endocrine, Neurological and Musculoskeletal systems) by the Investigator.
5. Subjects must be willing and able to attend all study visits and comply with "At-home" Instructions.
6. Subjects must be willing to have VISIA-CR facial photography imaging of their entire face for overall evaluation of their skin at all Visits.
7. Subjects must be willing and able to complete and understand the various rating questionnaires.
8. Subjects must have an IGA score of 2 (mild) or 3 (moderate) at the Baseline Visit.
9. Subjects must have a facial acne inflammatory lesion (papules, pustules, and nodules) count with no less than 10 but no more than 50 at the Baseline Visit.
10. Subjects must have a facial acne non-inflammatory lesion (open and closed comedones) count with no less than 10 but no more than 100 at the Baseline Visit.
11. Subjects with 1 or fewer facial nodules at the Baseline Visit.
12. Females of child bearing potential (FOCBP) and females who are premenses must be willing to practice effective contraception for the duration of the study. (Effective contraception is defined as stabilized on oral contraceptive for at least 3 months, intrauterine device, condom with spermicide, diaphragm with spermicide, implant, NuvaRing®, injection, transdermal patch or abstinence.) Females on birth control pills must have taken the same type pill for at least 3 months prior to entering the study and must not change type during the study. Those who have used birth control pills in the past must have discontinued usage at least 3 months prior to the start of the study. Women who use birth control for acne control only should be excluded.
13. Premenses females and FOCBP must have a negative urine pregnancy test at the Baseline Visit.
14. Subjects must be willing to comply with study instructions and return to the clinic for required visits.
15. Subjects must be willing to use the cleanser, moisturizer and sunscreen provided by the Sponsor.
16. If the subject wears makeup, they must agree to use non-comedogenic makeup.
17. Male subjects facial area must be clean-shaven for all study visits as to not interfere with study treatments and assessments.

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study.
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, Gram-negative folliculitis, dermatitis, eczema or an allergy to silicone.
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
4. Subjects with more than 50 facial acne inflammatory lesions (papules, pustules, and nodules)
5. Subjects with more than 100 facial acne non-inflammatory lesions (open and closed comedones)
6. Subjects with more than one (1) facial nodule.
7. Subjects with a facial beard or mustache that could interfere with the study treatments and assessments.
8. Subjects who have a history of experiencing significant burning or stinging when applying any facial treatment (e.g., makeup, soap, masks, washes, sunscreens, etc.) to their face.
9. Female subjects who are pregnant, nursing mothers, planning a pregnancy during the course of the study, or become pregnant during the study.
10. If female, subject has a history of hirsutism, polycystic ovarian disease or clinically significant menstrual irregularities.
11. Subjects who have a history of lupus erythematous, photosensitive eczema, albinism, photosensitive disorders (sensitization to light of the skin or eyes), light-induced seizures or diseases that may be stimulated by visible light.
12. Subjects currently using photosensitive medications or herbal supplements (see full list in Appendix IX) per the discretion of the Investigator assessment of risk.
13. Subjects who have a history of Herpes Simplex in the treatment area, connective tissue damage and immunosuppressive diseases.
14. Subjects who currently have active infections, broken skin, extremely dry skin or open lesions in the treatment area.
15. Treatment of any type of cancer within the last 6 months in the facial area, with the exception of complete surgical excision of skin cancer outside the treatment area.

18. Subjects who have not undergone the specified washout period(s) for the following topical preparations/physical treatments used on the face or subjects who require the concurrent use of any of the following in the treatment area:

Topical astringents and abrasives on the face 1 week Non-allowed moisturizers or sunscreens on the face 1 week Acne surgery 1 week Soaps containing antimicrobials on the face 1 week Antibiotics on the face 2 weeks Other topical anti-acne drugs on the face 2 weeks Chemical peel/Microdermabrasion on the face 2 weeks Light (PDT) therapy on the face 2 weeks Anti-inflammatory agents and corticosteroids on the face 4 weeks Retinoids, including retinol on the face 4 weeks Laser therapy on the face 4 weeks

19. Subjects who have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

Corticosteroids (including intramuscular injections) (inhaled corticosteroids are allowed) 4 weeks Antibiotics 4 weeks Other systemic acne treatments 4 weeks Systemic retinoids 6 months

20. Subject intends to use a tanning booth or sunbathe during the study. 21. Subjects who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

22. Subjects with any underlying disease that the investigator deems uncontrolled, and poses a concern for the subject's safety while participating in the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory lesion counts | Baseline to Day 49 or End of Study (EOS) visit
  Papule - A small, solid elevation less than 5 mm in diameter. Most of the lesion is above the surface of the skin.
  Pustule - A small circumscribed elevation less than 5 mm in diameter that contains yellow-white exudate.
  Nodule - An inflammatory lesion greater than or equal to 5 mm in diameter. Cyst - An inflammatory lesion that contains yellow-white exudate that is greater than or equal to 5mm in diameter.
Change in non-inflammatory lesion counts | Baseline to Day 49 or End of Study (EOS) visit
  Open Comedone - (Black head) A lesion in which the follicle opening is widely dilated with the contents protruding out onto the surface of the skin, with compacted melanin cells giving the plug a black appearance. Closed Comedone - (White head) A lesion in which the follicle opening is closed, but the sebaceous gland is enlarged by the pressure of the sebum buildup, which in turn cause the skin around the follicle to thin and become elevated with a white appearance.
Percentage/Proportion of subjects who achieve at least a one-grade reduction in the IGA Score | Baseline to Day 49 or End of Study (EOS) visit
  The Investigator will use the Investigator Global Assessment (IGA) Scale to assess the severity of a subjects' acne. The IGA Scale is a static evaluation should be performed prior to the lesion count. The IGA will be performed at Day 0, Day 21 and Day 49 or EOS. Subjects are eligible for enrollment if they have a global severity grade of a 2 (mild) or a 3 (moderate) on the IGA scale at Day 0. The following scores will be used to describe the severity grade:
  0 Clear Normal, clear skin with no evidence of acne vulgaris
  1. Almost Clear Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink red)
  2. Mild Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulo-cystic lesions)
  3. Moderate Multiple Non-inflammatory lesions and inflammatory lesions are evident, there may or may not be one small cyst
  4. Severe Inflammatory lesions are more apparent and a few cysts

SECONDARY OUTCOMES:
Improvement in Investigator Acne Scarring Assessment Scores using the Quantitative Global Acne Scarring Grading System (QGAS) | Baseline to Day 49 or End of Study (EOS) visit
  Patients' acne scarring will be evaluated by the Investigator using the Quantitative Global Acne Scarring Grading System (QGAS) as shown (Goodman and Baron, 2006). The QGAS will be performed at Baseline/Day 0, Day 21 and Day 49 or EOS. Only the face of the patient will be evaluated using the QGAS. This is a static morphological scale that refers to a point in time. The score will be calculated and recorded in the source.
  Milder scarring (1 point each) Macular erythematous or pigmented Mildly atrophic dish-like.
  Moderate scarring (2 points each) Moderately atrophic dish-like Punched out with shallow bases small scars (< 5 mm) Shallow but broad atrophic areas.
  Severe scarring (3 points each) Punched out with deep but normal bases, small scars (< 5 mm) Punched out with deep abnormal bases, small scars (< 5 mm) Linear or troughed dermal scarring Deep, broad atrophic areas Hyperplastic Papular scars (2 points each) Hyperplastic Keloid/hypertrophic scars (6 points each)
Improvement in Investigator Tolerability Assessment (erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation) | Baseline to Day 49 or End of Study (EOS) visit
  The scale is called Investigator Tolerability Assessment and the scale is 0 (None), 1 (Mild), (2) Moderate and 3 (Severe). The scale measures erythema, edema, dryness, scaling, hypopigmentation and hyperpigmentation. A decrease in scores (lower scores are a better outcome) or lack of significant increase at Day 21and Day 49 or EOS comparison to Baseline indicates tolerability/safety of the device.
Improvement in Acne QoL questionnaire scores | Baseline to Day 49 or End of Study (EOS) visit
  The Acne-specific Quality of Life questionnaire (Acne QoL) is a health-related quality of life instrument developed by MERCK & CO., INC. for use in clinical trials to assess the impact of therapy on quality of life among subjects with facial acne. The Acne QoL questionnaire consists of 19 questions. The Acne QoL is self-administrated (i.e. the subject is able to complete the questionnaire without assistance or interpretation from study staff) and should take approximately 10 minutes or less to complete. The scale is called Acne-Specific Quality of Life Questionnaire and the scale goes from 0 (not at all) to 6 (extremely). A decrease in response values (lower scores means a better outcome) at Day 49 or EOS indicates an improvement compared to baseline response values.
Improvement in Acne Self Assessment questionnaire scores | Baseline to Day 49 or End of Study (EOS) visit
  The Acne Self-Assessment Questionnaire will ask subjects a series of questions related to their facial acne and overall facial skin appearance. The scale is called the Acne Self-Assessment quesitonnaire and the scale goes from 0 (Very satisfied) to 5 (Very dissatisfied). A decrease in response values (lower scores means a better outcome) at Day 49 or EOS indicates an improvement compared to baseline response values.
Favorable Analysis of the Omnilux Clear® Device Subject Satisfaction questionnaire | Day 49 or EOS Visit
  The Omnilux Clear® Device Subject Satisfaction Questionnaire will ask subjects a series of questions related to their opinion of treatment satisfaction. The scale goes from 1 (Very Satisfied or Very Likely ) to 5 (Very Dissatisfied or Very Unlikely). Favorable analysis at Day 49 or EOS would be indicated by low response values.

OTHER OUTCOMES:
Improvement in the VISIA-CR photography imaging of the left, right and front views of the face. | Baseline to Day 49 or End of Study (EOS) visit
  Subjects will have VISIA-CR Facial imaging photographs taken of the right, central and left views of the face prior to Omnilux Clear treatment. All VISIA-CR facial images will be analyzed to acquire the following data points: (1) Visible Spots (2) Wrinkles (3) Texture (4) Pores (5) UV Spots (6) Brown Spots (7) Red Features (8) Porphyrins. The VISIA-CR software also formulates the following Ratings for Visible Spots, Wrinkles, Texture, Pores, UV Spots, Brown Spots, Red Features and Porphyrins:
  1. COUNT - The number of individual features detected within the region of interest (ROI) mask area.
  2. SCORE - The measure of feature severity. For the four spot algorithms (Visible Spots, UV Spots, Brown Spots and Red Features), score incorporates both fractional area and intensity. Otherwise, score is based only on fractional area. Measurement is normalized between 0 and 1. A lower score represents a lower amount of detection.
The frequency of both local and systemic AE's | Baseline, Day 21 and Day 49 or End of Study visit
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.
Subject Tolerability Self-Assessment (itching, burning and stinging) | Baseline, Day 21 and Day 49 or End of Study visit
  The scale is called Subject Tolerability Assessment and the scale is 0 (None), (1) Mild, (2) Moderate and 3 (Severe). The scale measures itching, burning and stinging. A decrease in scores (lower scores are a better outcome) or lack of significant increase at Day 21 and Day 49 or EOS comparison to Baseline indicates tolerability/safety of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Ablon Skin Institute and Research Center, Manhattan Beach, California, United States

IPD SHARING:
Plan to Share IPD: No